CLINICAL TRIAL: NCT02146690
Title: Effect of Osteopathic Manipulative Treatment on Reduction of Pain in Complicated Newborns: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Institute for Evidence Based Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEO-Pa 2
Record Dates: First submitted 2014-05-20; First posted 2014-05-26 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Prematurity
Keywords: pathology; newborn; osteopathic manipulative treatment; pain
MeSH Terms: conditions — Premature Birth; Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- osteopathic manipulative treatment (Other): newborns will receive osteopathic manipulative evaluation and treatment during the entire period of hospitalization plus usual care
  Interventions: Other: osteopathic manipulative treatment; Other: usual care
- sham (Other): newborns will receive sham treatment for the entire period of hospitalization plus usual care
  Interventions: Other: sham therapy; Other: usual care
- usual care (Other): newborns allocated in the usual care arm will receive standard care only
  Interventions: Other: usual care

INTERVENTIONS:
Other: osteopathic manipulative treatment
  Arms: osteopathic manipulative treatment
Other: sham therapy
  Arms: sham
Other: usual care

SUMMARY:
The aim of the present 3 armed placebo control parallel group randomized control trial is to explore the extent to which osteopathic manipulative treatment is effective in reducing pain in a population of complicated newborns.

ELIGIBILITY:
Inclusion Criteria:

* newborns born in the same hospital
* either gender
* diagnosis of any pathological/clinical medical condition

Exclusion Criteria:

* lack of guardian consent
* newborn transferred to/from other hospital
* lack of any of the inclusion criteria

Ages: 26 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-08 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
baseline changes in pain score using Premature Infant Pain Profile | baseline and end of hospitalization, expected hospitalization 4 weeks

SECONDARY OUTCOMES:
Length of stay in days | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

OTHER OUTCOMES:
Neonatal Intensive Care Unit cost | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Pescara Civil Hospital, Pescara, Italy